CLINICAL TRIAL: NCT04276337
Title: Genetic Characteristics of HER2 Positive Breast Cancer Receiving Neoadjuvant Chemotherapy With Docetaxel, Carboplatin, Trastuzumab and Pertuzumab (TCHP) Regimen
Brief Title: Genetic Characteristics of HER2 Positive Breast Cancer With Neoadjuvant TCHP Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, Professor, Samsung Medical Center
Other Study IDs: 2018-01-054
Record Dates: First submitted 2020-02-05; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: HER2-positive Breast Cancer; Chemotherapy Effect; Circulating Tumor DNA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood : circulating tumor DNA, Germline DNA Tissue : Targeted deep sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: LiquidSCAN(Trade Mark) / CancerSCAN(Trade Mark) — LiquidSCAN : detection of circulating DNA CancerSCAN : detection of somatic mutation using tumor tissue

SUMMARY:
Locally advanced breast cancer (LABC) is defined as breast cancer (BC) larger than 5 centimeters or with lymph node metastasis. Usually, LABC is treated with neoadjuvant chemotherapy (NAC) followed by curative surgery to reduce tumor size and eliminate micrometastasis. Response to NAC helps predict BC prognosis. Pathologic complete response (pCR), defined as no residual tumor cells after NAC, represents prolonged survival without BC recurrence and residual cancer burden score, based on residual tumor volume, and can more accurately predict BC outcomes. Especially, Human epidermal growth factor receptoor type 2(HER2)-positive breast cancer, having aggressive biologic characteristics, was mostly treated by NAC because of recent advance of highly effective targeted agents (pertuzumab and trastuzumab). However, still 30-40% of HER2-positive breast cancer did not response to NAC and underwent disease recurrence. Recently, genetic studies to find biomarker of BC prognosis have been widely performed. Circulating tumor DNA (ctDNA), which is circulating free DNA in the blood that originates from cancers, can be detected by recently-developed technologies. CtDNA could facilitate early disease detection, diagnosis and detection of disease recurrence. CtDNA also provides a genomic profile of BC and predicts drug response. In BC, ctDNA correlates with tumor burden and provides early detection of treatment response and tumor genetic alterations.

In this study, the investigator aimed to identify the correlations in genomic profile between tumors and ctDNA during NAC(docetaxel /carboplatin /trastuzumab and pertuzumab) in HER2 positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* HER2+ Breast cancer
* Stage IIA - IIIC
* Plan to receive neoadjuvant chemotherapy with docetaxel, carboplatin, herceptin, perjeta
* Sign to informed consent

Exclusion Criteria:

* Double primary cancer

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced HER2 positive breast cancer receiving neoadjuvant chemotherapy with docetaxel, carboplatin, trastuzumab and pertuzumab (TCHP) regimen
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response | Pathologic Clinical response is performed after end of cycle 6 (each cycle is 21 days)
  pCR of neoadjuvant(TCHP) chemotherapy with the patients with HER2 positive BC.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea